CLINICAL TRIAL: NCT01365507
Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec/Insulin Aspart Once Daily in Insulin-naïve Subjects With Type 2 Diabetes Mellitus When Using Two Different Titration Algorithms (BOOST™: SIMPLE USE)
Brief Title: Efficacy and Safety of Insulin Degludec/Insulin Aspart in Insulin-naïve Subjects With Type 2 Diabetes Using Two Dosing Regimens
Acronym: BOOST™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3844; U1111-1117-0558 (Other: WHO)
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp Simple (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IDegAsp Step wise (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Insulin degludec/insulin aspart injected subcutaneously (under the skin) once daily. Dose individually adjusted.
  Other Names: IDegAsp

SUMMARY:
This trial is conducted in Asia and North America. The aim of this trial is to compare the efficacy and safety of insulin degludec/insulin aspart (IDegAsp) once daily in insulin-naïve subjects with type 2 diabetes mellitus when using two different titration algorithms (dose individually adjusted) as add-on to subject's ongoing treatment with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for 24 weeks or longer prior to randomisation (visit 2)
* Insulin naïve subjects (Allowed are: Previous short term insulin treatment no longer than or equal to 14 days in total; Treatment during hospitalisation or during gestational diabetes is allowed for periods longer than 14 days in total)
* Current treatment: Metformin alone or metformin in any combination of 1 or 2 additional OADs (oral anti-diabetic drug) including an insulin secretagogue (sulfonylurea or glinide), dipeptidyl peptidase IV (DPP-IV) inhibitors, alpha-glucosidase inhibitors or thiazolidinediones (TZDs) - all with unchanged dosing for at least 12 weeks prior to randomisation (visit 2). Metformin dose, alone or in combination (including fixed combination), must be at least 1000 mg daily
* HbA1c (glycosylated haemoglobin) 7.0-10.0% (both inclusive)
* BMI (Body Mass Index) below or equal to 45 kg/m^2
* Ability and willingness to adhere to the protocol including self measurement of plasma glucose

Exclusion Criteria:

* Treatment with GLP-1 (glucagon like peptide) receptor agonists within the last 12 weeks prior to randomisation (visit 2)
* Recurrent severe hypoglycaemia (more than one severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator (trial physician)
* Previous participation in this trial. Participation is defined as randomised. Re-screening is allowed once during the recruitment period
* Known or suspected hypersensitivity to trial products or related products
* The receipt of any investigational drug within 4 weeks prior to randomisation (visit 2)
* Anticipated significant lifestyle changes during the study, e.g. shift work (including permanent night/evening shift workers) as well as highly variable eating habits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (35):
- United States (23):
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Crestview Hills, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, North East, Maryland
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Eagan, Minnesota
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Malaysia (3):
  - Novo Nordisk Investigational Site, Johor Bahru
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Kuala Selangor
- Mexico (2):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Monterrey
- Novo Nordisk Investigational Site, Bayamón, Puerto Rico
- South Korea (2):
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
- Thailand (2):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Nakhon Ratchasima
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul

REFERENCES:
- [Result] Park SW, Bebakar WM, Hernandez PG, Macura S, Herslov ML, de la Rosa R. Insulin degludec/insulin aspart once daily in Type 2 diabetes: a comparison of simple or stepwise titration algorithms (BOOST(R) : SIMPLE USE). Diabet Med. 2017 Feb;34(2):174-179. doi: 10.1111/dme.13069. Epub 2016 Mar 6. PMID 26773557
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 38 sites in 6 countries: Malaysia, Mexico, South Korea, Thailand, Turkey and the United States (U.S.).
Pre-assignment Details: Subjects continued their metformin monotherapy or metformin in any combination with 1 or 2 additional oral antidiabetic drugs including an insulin secretagogue (sulfonylurea or glinide), dipeptidyl peptidase IV inhibitors, α-glucosidase inhibitors, thiazolidinediones, all with unchanged dosing for at least 12 weeks prior to randomisation.
Groups:
- IDegAsp Simple: Insulin degludec/insulin aspart (IDegAsp) was given once daily (OD) subcutaneously (3-4 days intervals between doses) with pre-trial metformin according to simple titration algorithm: self-titration was performed twice weekly based on pre-breakfast self-measured plasma glucose (SMPG) value measured on the day of insulin titration.
- IDegAsp Step Wise: Insulin degludec/insulin aspart (IDegAsp) was given once daily (OD) subcutaneously (at least 5 days intervals between doses) with pre-trial metformin according to step wise titration algorithm: self-titration was performed once weekly based on the lowest value of three pre-breakfast SMPG values measured on three consecutive days, the two days prior to and on the day of insulin titration.
Period: Overall Study
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Started | 136 | 140
Exposed | 134 (Two subjects withdrew before exposure to trial drug) | 140
Completed | 127 | 131
Not Completed | 9 | 9
Not completed — Withdrawal Criteria | 8 | 5
Not completed — Unclassified | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp Simple | IDegAsp Step Wise | Total
Number analyzed (Participants) | 136 | 140 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.4) | 55.8 (9.7) | 56.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 84 | 143
  Male | 77 | 56 | 133
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.8) | 8.2 (0.8) | 8.3 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.9 (2.4) | 9.0 (2.3) | 8.9 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 136 | 140
percentage of glycosylated haemoglobin | -1.33 (1.03) | -1.09 (0.82)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). For 2 subjects baseline values were missing, hence not included in the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 135 | 139
mmol/L | -2.99 (3.03) | -2.73 (2.91)

3. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 134 | 140
Events/100 years of patient exposure
  Adverse events (AEs) | 226 | 342
  Serious AEs | 2 | 13
  Severe AEs | 3 | 3
  Moderate AEs | 68 | 112
  Mild AEs | 155 | 228
  Fatal AEs | 0 | 0

4. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 134 | 140
Episodes/100 years of patient exposure | 326 | 207

5. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of nocturnal confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes were defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 134 | 140
Episodes/100 years of patient exposure | 52 | 41

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up.
Description: The safety analysis set included all subjects who received at least one dose of the investigational product.
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Serious Adverse Events (participants affected / at risk) | 1/134 | 6/140
Other Adverse Events (participants affected / at risk) | 20/134 | 26/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp Simple (N=134) | IDegAsp Step Wise (N=140)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp Simple (N=134) | IDegAsp Step Wise (N=140)
Nasopharyngitis (Infections and infestations) | 8 (10) | 11 (13)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.